CLINICAL TRIAL: NCT04415866
Title: Generalized Hypersensitivity in Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202000992
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: central sensitization; peripheral sensitization; visual evoke potentials (VEP); quantitative sensory testing
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Participants sensitivity to pressure, heat, and light will be modulated by an attention task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of PASAT on Sensory Testing (Experimental): After baseline evaluation of light and pain sensitivity FM subjects and controls will undergo the PASAT task. This task consists of responding to a rapid presentation of numbers by ear phones. Subjects are asked to add each 2 consecutive numbers and provide a response each time the sum is equal to 13. This test will last several minutes and delivered at increasing speed.
  Interventions: Behavioral: Paced Auditory Serial Addition task (PASAT)

INTERVENTIONS:
Behavioral: Paced Auditory Serial Addition task (PASAT) — Single and double digits are presented at intervals between 2 and 3 seconds and the participant must add each new digit to the one immediately prior to it. The participants will be asked to indicate by electronic button press whether the sum of the addition is 13 or not. The duration of the PASAT will be two 12-min tasks.

SUMMARY:
Fibromyalgia (FM) is a chronic musculoskeletal pain disorder with unknown causes. Our previous studies showed abnormal sensations of second pain (wind-up), indicating central hypersensitivity as an important mechanism of FM. Triggering events have been implicated as the cause of central hypersensitivity.

DETAILED DESCRIPTION:
Increasing evidence has shown that the hypersensitivity of FM is not limited to painful stimuli but seems to extend to non-painful stimuli as well. These stimuli include smell, taste, touch, light, and sound. This study will provide detailed QST examinations of FM subjects and controls' responses to light using visually evoked potentials (VEP). In addition, careful characterization of experimental pain responding across multiple sensory modalities will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with FM will have pain of > 3 months and meet the 1990 and 2011 Diagnostic Criteria for FM (ACR)
* Healthy, pain-free age and sex matched controls without chronic pain

Exclusion Criteria:

* Presence of chronic disease (e.g. cancer, cardiovascular disease, liver disease, kidney disease, diabetes, etc.).
* FM patients must be willing to discontinue or hold their FM related medications for a minimum of one day prior to the visit.
* Significant vision loss not corrected by eye wear
* Family history of photosensitive epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Verbal Pain Ratings of Painful Heat and Pressure Stimuli using a Numerical Pain Scale from 0 - 100 | 1 hour
  FM and control subjects will provide verbal ratings of experimental pain stimuli. For this purpose a numerical ratings scale (0-100) will be used ranging from "no sensation" to the "most intense sensation possible". All measures will be obtained in triplicates and the averages will be used for statistical comparisons.
Visual Evoked Potentials (VEP) During Flicker | 1 hour
  FM and control subject will focus on a light source while VEPs are obtained. EEG tracings will be evaluated by special software to detect VEP. For intensity ratings of the flicker stimulus a numerical ratings scale (0-100) will be used ranging from "no sensation" to the "most intense sensation possible". All measures will be obtained in triplicates and the averages will be used for statistical comparisons.

SECONDARY OUTCOMES:
Response to 2011 Fibromyalgia Criteria Questionnaire | 0.5 hours
  FM and control subjects will complete the 2011 FM Questionnaire. The answers of this questionnaire will be added to obtain the wide-spread pain index and the somatic symptom score. The scores will be combined to obtain the final score. Scores of >12 fulfill the Criteria for Fibromyalgia
Response to the Center for Epidemiological Studies (CES-D) Depression Questionnaire | 0.5 hours
  FM and control subjects will complete the CES-D. The answers of this questionnaire will be combined to obtain a final score. Total scores of >15 are consistent with the diagnosis of major depression.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geisser ME, Strader Donnell C, Petzke F, Gracely RH, Clauw DJ, Williams DA. Comorbid somatic symptoms and functional status in patients with fibromyalgia and chronic fatigue syndrome: sensory amplification as a common mechanism. Psychosomatics. 2008 May-Jun;49(3):235-42. doi: 10.1176/appi.psy.49.3.235. PMID 18448779
- [Background] Geisser ME, Glass JM, Rajcevska LD, Clauw DJ, Williams DA, Kileny PR, Gracely RH. A psychophysical study of auditory and pressure sensitivity in patients with fibromyalgia and healthy controls. J Pain. 2008 May;9(5):417-22. doi: 10.1016/j.jpain.2007.12.006. Epub 2008 Feb 15. PMID 18280211
- [Background] Frank MG, Fonken LK, Watkins LR, Maier SF. Microglia: Neuroimmune-sensors of stress. Semin Cell Dev Biol. 2019 Oct;94:176-185. doi: 10.1016/j.semcdb.2019.01.001. Epub 2019 Jan 9. PMID 30638704
- [Background] Geisser ME, Casey KL, Brucksch CB, Ribbens CM, Appleton BB, Crofford LJ. Perception of noxious and innocuous heat stimulation among healthy women and women with fibromyalgia: association with mood, somatic focus, and catastrophizing. Pain. 2003 Apr;102(3):243-250. doi: 10.1016/S0304-3959(02)00417-7. PMID 12670665